CLINICAL TRIAL: NCT05906667
Title: Sharing History Through Active Reminiscence and Photo-imagery: A Neighborhood Approach to Increase Physical Activity and Social Engagement
Brief Title: Sharing History Through Active Reminiscence and Photo-imagery - With MCI
Acronym: SHARP-MCI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00016980
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: single-arm study; all participants are assigned to the experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All participants assigned to the experimental group (walking)
  Interventions: Behavioral: Sharing History through Active Reminiscence and Photo-imagery (SHARP)

INTERVENTIONS:
Behavioral: Sharing History through Active Reminiscence and Photo-imagery (SHARP) — Participants engage in neighborhood walks and conversational reminisce three times per week over 24 weeks
  Other Names: SHARP

SUMMARY:
The SHARP-MCI study tests impact of walking and social reminiscence on cognitive function, blood pressure, and weight among healthy Black Americans and those experiencing mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
For 6 months (24 weeks), triads of healthy and MCI Black adults aged 55 and over walk 3x/week (1 mile) in Portland's historically Black neighborhoods. Triads follow GPS-mapped routes accessible via the SHARP walking application on a group tablet device. At three points along each route, GPS-triggered "Memory Markers" (historical images of local Black culture and life from1940-2010) appear on the tablet screen serving as a conversational reminisce prompt as the triad walks. At baseline and 24 weeks, cognitive function is measured via the Montreal Cognitive Assessment (MoCA), and weight and blood pressure are measured. Pre-post health surveys rate activity levels, days feeling downhearted/blue, energy level, and health status. Program evaluation surveys at month 1, 3, 6 assess mood, pace and dose of walking, prompt effectiveness, program readiness, and liklihood to recommend program to others. Focus groups at month 1, 3, 6 evaluate participants' program experience and needed changes.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American
* > 55 years old
* Reside or resided for >10 years in Portland's historically Black neighborhoods (to be familiar with Memory Markers about this area)
* Able to ambulate independently. Participants (n=7) with MCI will meet criteria consistent with those defined by Jak et al. 2009 and with criteria outlined by the NIA-Alzheimer's Association workgroup (2011)
* Participants without cognitive impairment (n=14) will have an MMSE score > 24 (and not meet MCI criteria).
* Participants' cognitive function should allow them to get to/ from walk locations independently or with minimal assistance

Exclusion Criteria:

* Serious or unstable medical condition (such as, but not limited to, cardiovascular disease, pulmonary disease, or severe arthritis) where participation in the trial would, in the opinion of the investigator, pose a significant health risk to the subject.
* Diagnosis of Alzheimer's disease, vascular dementia, Parkinson's disease, or other dementing illness.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 24 weeks
  Pre/post Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Blood pressure | 24 weeks
  pre/post blood pressure reading
Weight | 24 weeks
  pre/post weight measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carder, P., Croff, R., Tuttle, A., Towns, J. (2022) Walking and Talking: Recommendations for Doing Mobile Interviews with Older Adults. Journal of Aging and Environment, DOI: 10.1080/26892618.2022.2030844
- [Derived] Croff R, Aron S, Wachana A, Fuller P, Mattek N, Towns J, Kaye J. Walking and Social Reminiscence in Gentrifying Neighborhoods: Feasibility and Impact on Cognitive, Physical, and Mental Health Among Older Black Adults in the SHARP Study. Gerontologist. 2024 Sep 1;64(9):gnae019. doi: 10.1093/geront/gnae019. PMID 38412543